CLINICAL TRIAL: NCT05635162
Title: Zanubrutinib Plus Rituximab (Zanu -R) as Fixed Duration, Early Intervention Versus Observation for Patients With Indolent Mantle Cell Lymphoma: a Randomised Phase II Clinical Trial
Brief Title: Zanubrutinib Plus Rituximab for Patients With Indolent Mantle Cell Lymphoma
Acronym: ZEBRA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL 146660
Record Dates: First submitted 2022-10-31; First posted 2022-12-02 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — zanubrutinib; Rituximab

STUDY DESIGN:
Intervention Model Description: Randomised
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Control (No Intervention): Active observation
- Arm B: Experimental (Experimental): Time limited Zanubrutinib-R 6 x 28 day cycles
  Interventions: Drug: Zanubrutinib; Drug: Rituximab

INTERVENTIONS:
Drug: Zanubrutinib — Zanubrutinib dose is 160 mg twice daily (BD) orally (PO) on days 1-28 of each 28-day cycle.
  Arms: Arm B: Experimental
Drug: Rituximab — Rituximab 375 mg/m2 intravenous (IV)* on day 1 (+/-3 days) of each 28-day cycle
  Arms: Arm B: Experimental

SUMMARY:
Phase II, multicentre, randomised, open-label study to assess the benefit of early intervention with fixed duration, time-limited zanubrutinib-rituximab in indolent mantle cell lymphoma (MCL)

DETAILED DESCRIPTION:
This is a phase II, multicentre, randomised open label study to assess the safety and efficacy of zanubrutinib in combination with rituximab for previously untreated indolent MCL patients.

50 patients will be recruited from 15 UK centres over 30 months.

Enrolled patients will be randomised (1:1) to ongoing observation (control arm; arm A) or fixed-duration zanubrutinib-rituximab (experimental arm; arm B). Patients will discontinue zanubrutinib-rituximab after 6 cycles of therapy or sooner in the advent of unacceptable toxicity or any other reason.

All patients will be followed up for a minimum of 2 years after randomisation. Patients in arm B who develop disease progression and require further therapy after the initial time-limited Zanu-R will receive standard of care therapy according to front line treatment available at that time.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or over.
2. Life expectancy ≥ 6 months.
3. Pathologically confirmed MCL, with documentation of monoclonal B cells that have a chromosome translocation t(11;14)(q13;q32) and/or overexpress cyclin D1, D2 or D3.
4. Stage II-IV MCL measurable by CT imaging or by white cell count (WCC)/BM infiltration.
5. 'Indolent' MCL, defined as 1 or more of the following:

   * Observation with no treatment for a minimum of 6 months after the initial diagnosis
   * Leukaemic non-nodal variant (lymphocytosis/splenomegaly only without nodal involvement)
   * Low tumour volume (largest lymph node ≤ 3cm in maximal diameter), proliferation fraction (Ki67 or equivalent) ≤30% and classical morphology (non-blastoid/pleomorphic)
6. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2.
7. Absolute neutrophil count ≥1.0 x 109/L and platelets ≥75 x 109/L independent of growth factor support.
8. AST and/or ALT ≤3 x upper limit of normal (ULN).
9. Total Bilirubin ≤1.5 x ULN unless due to Gilberts syndrome or of non-hepatic origin unless directly attributable to the patient's MCL.
10. Calculated creatinine clearance ≥30 mL/min. Glomerular filtration rate (GFR) ≥30 mL/min directly measured with 24 hour urine collection, or creatinine clearance calculated according to the modified formula of Cockcroft and Gault (for men: GFR ≈ ((140 - age) x bodyweight)/ (72 x creatinine), for women x 0, 85).
11. Able to give voluntary written informed consent.
12. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty.
13. Negative serum or urine pregnancy test for women of childbearing potential (WOCBP).
14. Willing to comply with the contraceptive requirements of the trial.

Exclusion Criteria:

1. Any prior therapy for MCL, including prior radiotherapy.
2. Central nervous system (CNS) involvement of MCL.
3. Uncontrolled infection with HIV or any uncontrolled active systemic infection (e.g., bacterial, viral or fungal). Patients with well-controlled HIV status (undetectable viral load) will not be excluded.
4. Hepatitis B or C serologic status: subjects who are hepatitis B core antibody (anti-HB core) positive and who are surface antigen (HBsAg) negative will need to have a negative polymerase chain reaction (PCR) test. Those who are hepatitis B HbsAg positive or hepatitis B PCR positive will be excluded. Those who are hepatitis C antibody and PCR positive will be excluded (those who are hepatitis C antibody positive and PCR negative will not be excluded).
5. No progression requiring treatment since initial diagnosis.
6. Vaccinated with live vaccines (not including messenger ribonucleic acid (mRNA), viral vector or other non-live COVID19 vaccines) within four weeks prior to randomisation.
7. Major surgical procedure within 28 days prior to randomisation. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
8. Prior malignancy (or any other malignancy requiring active treatment), except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, localised prostate cancer or other cancer from which the subject has been disease free for ≥ 2 years or which will not limit survival to < 5 years.
9. Requirement for moderate or strong CYP3A inducers. Moderate and strong CYP3A inhibitors are allowed although these should be switched to agents causing less CYP3A inhibition where possible.
10. Requirement for vitamin K antagonists (alternative anticoagulation is allowed (e.g. DOACs), but patients must be properly informed about the potential risk of bleeding alongside zanubrutinib). Requires ongoing treatment with warfarin or warfarin derivatives
11. Active bleeding or history of bleeding diathesis (e.g. haemophilia or von Willebrand disease) or history of spontaneous bleeding requiring blood transfusion or other medical intervention.
12. Clinically significant cardiovascular disease such as uncontrolled arrhythmias, or history of ventricular tachycardia, ventricular fibrillation, torsades de points or myocardial infarction within 6 months of randomisation, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association (NYHA) Functional Classification, or corrected QT interval (QTc) > 480 msec, second-degree atrioventricular block Type II, third-degree atrioventricular block at randomisation, unstable angina within 3 months prior to randomisation.
13. History of stroke or intracranial haemorrhage within 6 months prior to randomisation.
14. Any other severe medical or psychiatric illness that in the opinion of the investigator would interfere with participation in this clinical study.
15. Malabsorption syndrome, unable to swallow capsules, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
16. Women who are pregnant or breastfeeding.
17. Male participants with female partners of childbearing potential who are unwilling to use appropriate contraception methods.
18. Concurrent treatment with another investigational agent.
19. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies, known sensitivity or allergy to murine products.
20. Known hypersensitivity to any active substance or to any of the excipients of one of the drugs used in the trial.
21. Severe or debilitating pulmonary disease.
22. Underlying medical conditions that, in the investigator's opinion, will render the administration of study drug hazardous or obscure the interpretation of toxicity or AEs
23. Concurrent participation in another therapeutic clinical trial.
24. Active and/or ongoing autoimmune anaemia and/or autoimmune thrombocytopenia (eg. idiopathic thrombocytopenia purpura).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-17 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Event free survival | From date of randomisation until whichever comes first: occurrence of active disease, new MCL treatment or death (any cause) up to 60 months
  To determine the effect of fixed-duration Zanu-R on Event-free survival (EFS) compared to active observation

SECONDARY OUTCOMES:
Progression free survival | Randomisation until disease progression up to 60 months
  To determine the effect of fixed-duration Zanu-R on Progression free survival (PFS) compared to active observation
Overall survival | Randomisation until date of death up to 60 months
  To determine the effect of fixed-duration Zanu-R on overall survival (OS) compared to active observation
Time to next treatment | Randomisation until date of initiation of subsequent treatment up to 60 months
  To determine the effect of fixed-duration Zanu-R on time to next treatment (TTNT) compared to active observation
Time to second progression | From date of randomisation or date of first progression until date of second progression or death from any cause up to 60 months
  To determine the effect of fixed-duration Zanu-R on time to second progression compared to active observation
Overall response rate to Zanu-R | From start of treatment until 24 weeks post administration of Zanu-R
  To determine the effect of fixed-duration Zanu-R on overall response rate (ORR) at the end of 6 cycles of treatment
Overall response rate to re-treatment with covalent BTKi | From the start of further treatment with a BTKi through to study completion, an average of 60 months
  To determine the ORR to re-treatment with covalent BTKi in experimental arm
Safety and Toxicity | From informed consent until 28 weeks post randomisation
  To assess the worst grade of each adverse event for each patient. Grades 1-2 and grades 3-5 will be compared between the arms

CONTACTS AND LOCATIONS:
Locations (13):
- United Kingdom (13):
  - Royal Derby Hospital, Derby
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Clatterbridge Cancer Centre, Liverpool
  - Guy's Hospital, London
  - St Bartholomew's Hospital, London
  - University College London Hospital, London
  - Christie Hospital, Manchester
  - Norfolk and Norwich University Hospitl, Norwich
  - Nottingham City Hospital, Nottingham
  - Churchill Hospital, Oxford
  - Derriford Hospital, Plymouth
  - Southampton General Hospital, Southampton
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: Undecided